CLINICAL TRIAL: NCT01046825
Title: Mature B-Cell Lymphoma And Leukemia Study III
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJBC3; NCI-2011-01251 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2025-05-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Mature B-Cell Lymphoma
Keywords: Lymphoma; Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma; Leukemia; Lymphoma, Non-Hodgkin | interventions — Prednisone; Doxorubicin; Cyclophosphamide; Filgrastim; pegfilgrastim; rasburicase; Leucovorin; Rituximab; Cytarabine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Other): Completely resected stage I or completely resected abdominal stage II lesions.
  Group A will include: COPAD x 2 cycles.
  Interventions: Drug: COPAD
- Group B (Other): All cases not eligible for Group A or Group C. (Murphy Stage III and non-CNS Stage IV)
  Group B will include the intervention COP, COPD M3, CYM as follows:
  Pre-Phase: COP
  Induction: COPAD M3 x 2 cycles
  Consolidation: CYM x 2 cycles.
  Interventions: Drug: COP, COPD M3, CYM
- Group C (Other): Any CNS involvement and/or bone marrow involvement ≥ 25% blasts. For CNS involvement one or more of the following applies:
  1. Any L3 blasts in CSF
  2. Cranial nerve palsy (if not explained by extracranial tumor)
  3. Clinical spinal cord compression
  4. Isolated intracerebral mass
  5. Parameningeal extension: cranial and/or spinal
  Group C will include the intervention COP, COPADM8, CYVE as follows:
  Pre-Phase: COP
  Induction: COPADM8 cycle 1
  Induction: COPADM8 Cycle 2
  Consolidation: CYVE x 2 cycles
  and Maintenance
  Interventions: Drug: COP, COPADM8, CYVE

INTERVENTIONS:
Drug: COPAD — Vincristine Prednis(ol)one, Cyclophosphamide, Doxorubicin, G-CSF
  In the event the patient cannot receive G-CSF, Pegfilgrastim can be substituted.
  Other Names: VCR; prednisone; Adriamycin; cytoxan; filgrastim; Neupogen; Neulasta®
  Arms: Group A
Drug: COP, COPD M3, CYM — GROUP B Treatment Details Intravenous fluids should be given at a rate of 3000 mL/m2/day. Use of rasburicase may preclude the need for HCO3 Pre-Phase: Cyclophosphamide, Vincristine, Prednis(ol)one, IT medications Induction (2 cycles): Vincristine, Prednis(ol)one, Methotrexate, Leucovorin, Cyclophosphamide, Doxorubicin, IT medications, G-CSF, Rituximab Consolidation (2 cycles): Methotrexate, Leucovorin, Cytarabine, IT medications, G-CSF, Rituximab
  In the event the patient cannot receive G-CSF, Pegfilgrastim can be substituted.
  Other Names: Elitek; Cytoxan; VCR; prednisone; MTX; folinic acid; Adriamycin; filgrastim; Rituxan; Ara-C; Neulasta®
  Arms: Group B
Drug: COP, COPADM8, CYVE — Treatment: Intravenous fluids should be given at a rate of 3000 mL/m2/day. Use of rasburicase may preclude the need for HCO3.
  COP Pre-Phase: Cyclophosphamide, Vincristine, Prednis(ol)one, IT medications, Leucovorin.
  COPADM8 Induction (2 cycles): Vincristine, Prednis(ol)one, Methotrexate, Leucovorin, Cyclophosphamide, Doxorubicin, Rituximab, IT medications, G-CSF CYVE Consolidation (2 cycles): Cytarabine, High-Dose Ara-C, Etoposide, Rituximab, G-CSF.
  Maintenance No.1: Vincristine, Prednis(ol)one, Cyclophosphamide, Methotrexate, Leucovorin, Doxorubicin, IT medications, G-CSF.
  Maintenance No.2: Cytarabine, Etoposide, G-CSF, IT Medications. Maintenance No.3: Vincristine, Prednis(ol)one, Cyclophosphamide, Doxorubicin, G-CSF, IT Medications.
  Maintenance No. 4: Cytarabine, Etoposide, G-CSF, IT Medications.
  In the event the patient cannot receive G-CSF, Pegfilgrastim can be substituted.
  Other Names: Elitek; cytoxan; VCR; prednisone; folinic acid; Adriamycin; filgrastim; Ara-C; VP16; MTX; Rituxan; Neulasta®
  Arms: Group C

SUMMARY:
This is a phase III clinical trial using risk-adapted therapy. Treatment outcomes for children with B-cell NHL are excellent. Further improvements in outcome will likely be achieved through more focused study of the biology of the tumors and prospective studies of the late effects of treatment. Toward this end, this study features a spectrum of prospective biologic and late effect studies performed in patients treated with a modified regimen derived from the very successful LMB-96 regimen.

DETAILED DESCRIPTION:
1. This study will perform analysis of newly diagnosed mature B-cell lymphomas (e.g. Burkitt lymphoma/leukemia, DLBCL, and MLBCL) obtained from participants in different parts of the world.
2. This study will describe the types and frequency of mutations in the ARF-HDM2-TP53 pathway, in B-cell lymphomas in the United States and that found in selected geographic regions of the world.
3. This study will describe the expression of ARF-HDM2-TP53 and PUMA-associated pathways in B-cell lymphomas in the United States and that found in B-cell lymphomas of other selected geographic regions of the world.
4. This study will describe the pattern and frequency of XLP gene mutations presenting with B-cell lymphomas in the United States and selected geographic regions.
5. This study will describe the frequency of EBV-positive B-cell lymphomas in the United States and selected geographic regions of the world: and will describe the pattern of EBV protein and gene expression (e.g., EBNA 3) in EBV-positive lymphomas and the study will compare patterns of EBV protein and gene expression with clinical, laboratory and outcome data.

Exploratory Aims:

To estimate the complete response rate, event-free survival, and overall survival rates in patients with Burkitt lymphoma (BL), Burkitt leukemia/B-cell acute leukemia (B-ALL) and diffuse large B-cell lymphoma (DLBCL) treated with a stage-adapted regimen based on the St. Jude B-cell II protocol.

ELIGIBILITY:
Inclusion Criteria:

St. Jude participants and collaborating sites participating in therapeutic and biological objectives:

1. Participant must have a histologic diagnosis of a mature B cell lymphoma (e.g., Burkitt lymphoma/leukemia, atypical Burkitt lymphoma, diffuse large B-cell lymphoma, mediastinal large B-cell lymphoma, mature B-cell lymphoma NOS) as defined in the WHO classification.
2. Participant must be previously untreated, (no more than 72 hours of steroids, one intrathecal chemotherapy treatment, and/or emergency radiation).
3. Participant must be < 22 years of age at the time of diagnosis
4. For selected higher-risk CD20+ Group B and all CD20+ Group C participants receiving rituximab only (e.g., those with MLBLC, Stage III with LDH ≥ 2 times upper limit of normal (ULN), and/or bone marrow/CNS involvement: All participants who will receive rituximab must have hepatitis screening prior to enrollment. Participants whose results indicate that they are carrier of hepatitis B can still be treated per Group B or C but will NOT receive rituximab. This screening must be done for eligibility for participants who will receive rituximab, BUT the results are not needed prior to enrollment:

   * Hepatitis B immunization status (vaccination Yes or No)
   * HBsAg
   * Anti-HBs antibody
   * Anti-HBc antibody.
5. All participants must have screening prior to enrollment; participants whose results indicate that they are carrier of hepatitis B can still be treated per group B and C but will NOT receive rituximab
6. HIV test has been obtained within 42 days. Participants who test positive for HIV cannot be enrolled on therapeutic part of study, but are still eligible for biology studies.
7. Informed consent must be obtained according to St. Jude guidelines before enrollment into study.

Participants from Collaborating Sites Participating in Biological Objectives Only:

1. Participant must have a histologic diagnosis of a mature B cell lymphoma (e.g., Burkitt lymphoma/leukemia, atypical Burkitt lymphoma, diffuse large B-cell lymphoma, mediastinal large B-cell lymphoma, mature B-cell lymphoma NOS) as defined in the WHO classification.
2. Participant must be < 22 years of age at the time of diagnosis.
3. Participant must be previously untreated (no more than 72 hours of steroids, one intrathecal chemotherapy treatment, and/or emergency radiation) at the time of the diagnostic biopsy.
4. Informed consent must be obtained by local PI or his/her designee according to ICH/Good Clinical Practice and local guidelines before enrollment into study.

Exclusion Criteria:

Participants from Collaborating Sites Participating in Therapeutic and Biological Objectives:

1. Participants known to be HIV positive (for therapeutic part of protocol, HIV participants are eligible for biology studies).
2. Participants who are pregnant or lactating.
3. Inability or unwillingness of research participant or legal guardian to consent.

Participants from Collaborating Sites Participating in Biological Objectives Only:

1. Inability or unwillingness of research participant or legal guardian to consent.
2. Histologic diagnosis other than a mature B-cell lymphoma as defined in the WHO classification.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2027-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Ribeiro, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (2):
  - Rady Children's Hospital San Diego, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Children's Cancer Hospital, Cairo, Egypt
- National University Health System, Singapore, Singapore

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 patients were recruited between 15APR1309Sept2010 and 31AUG2022. One patient died at the same day he was enrolled and did not start any treatment and risk was not determined and was excluded in the treatment outcome analysis. One was found to be ineligible after the start of treatment.
  Thirteen participants from diverse geographical regions were enrolled in the biology only part of the study and no outcome data is available.
Groups:
- Group A: Completely resected stage I or completely resected abdominal stage II lesions.
- Group B: All cases not eligible for Group A or Group C. (Murphy Stage III and non-CNS Stage IV)
- Group C: Any CNS involvement and/or bone marrow involvement ≥ 25% blasts. For CNS involvement one or more of the following applies:
  1. Any L3 blasts in CSF
  2. Cranial nerve palsy (if not explained by extracranial tumor)
  3. Clinical spinal cord compression
  4. Isolated intracerebral mass
  5. Parameningeal extension: cranial and/or spinal
- Unknown Risk: Patient died prior to treatment and risk assignment
- Biology Only: Participants enrolled on the biology only arm
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Unknown Risk | Biology Only
Started | 5 | 87 | 22 | 1 | 13
Completed | 5 | 84 | 19 | 0 | 0
Not Completed | 0 | 3 | 3 | 1 | 13
Not completed — Failed to achieve CR to Induction Therapy | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0
Not completed — Participant or family decision to withdraw from protocol treatment | 0 | 0 | 1 | 0 | 0
Not completed — Found to be ineligible | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Did not submit biology samples | 0 | 0 | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Of the 87 participants that started in Group B, one was found to be ineligible and is excluded from all analysis, including adverse events.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Biology Only | Total
Number analyzed (Participants) | 5 | 86 | 22 | 13 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (4.1) | 12.4 (5.1) | 13.0 (5.5) | 13.4 (5.8) | 12.5 (5.1)
Age, Continuous [Median (Full Range); unit: years] | 13.7 [8.01 to 18.7] | 12.9 [3.0 to 20.8] | 14.4 [2.5 to 20.9] | 14.7 [3.8 to 24.8] | 13.4 [2.5 to 20.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 21 | 7 | 2 | 32
  Male | 3 | 65 | 15 | 11 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 64 | 18 | 1 | 87
  Black | 0 | 12 | 4 | 0 | 16
  Asian | 1 | 4 | 0 | 11 | 16
  Multiple Race (Not Otherwise Specified) | 0 | 4 | 0 | 0 | 4
  Other | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Gene Differential Expression Profiling of Burkitt Lymphoma (BL) vs. Non-BL in the US and Other Selected Geographic Regions of the World
Description: Gene expression levels in BL vs. non-BL will be analyzed through approximately 22,000 probesets on the Affymetrix U133A GeneChip by using two-factor analysis of variance model for each gene.
Time Frame: 1 year after the participant is enrolled
Population: No data was generated for this measure due to the PI leaving St. Jude, COVID-19 disruptions, stricter regulations on international tumor material shipping, and unavailability of the required assay platform. One sample was received from Singapore, none from Egypt. No participant is analyzed, and no gene expression data is generated because the Affymetrix U133A GeneChip is no longer available. No participant will be analyzed, and no gene expression data will be generated in the future.
Groups:
- Biology Samples-United States (US): US Participants Biology Samples
- Biology Samples-Singapore: Singapore Participants Biology Samples
- Biology Samples-Egypt: Egypt Participants Biology Samples
Arm/Group | Biology Samples-United States (US) | Biology Samples-Singapore | Biology Samples-Egypt
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Catalog and Estimate Frequencies of Copy Number Variations in Childhood Lymphomas
Description: The prevalence of CNVs between different subtypes of childhood lymphomas and geographic regions will be reported and compared with exact chi-square or Fisher's test. The CNVs are derived from Affymetrix SNP arrays.
Time Frame: 1 year after the participant is enrolled
Population: We were unable to evaluate this measure due to challenges such as the PI leaving St. Jude, COVID-19 disruptions, stricter regulations on shipping tumor materials internationally, and unavailability of the required assay platform. One sample was received from Singapore, none from Egypt. No participant is analyzed, and no CNV data is generated because the Affymetrix SNPChip platform is no longer available. No participant will be analyzed, and no CNV data will be generated in the future.
Arm/Group | Biology Samples-United States (US) | Biology Samples-Singapore | Biology Samples-Egypt
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Integrated Analysis of CNVs and Gene Expressions in the US and Other Selected Geographic Regions of the World
Description: The association between the identified CNVs and gene expressions in the study cohort will be examined by using general linear models, and multiple tests will be considered. Gene expressions are measured by Affymetrix U133A arrays and CNVs are derived from Affymetrix SNP arrays.
Time Frame: 1 year after the participant is enrolled
Population: No data was generated for this measure due to PI leaving St. Jude, COVID-19 disruptions, stricter regulations on international tumor material shipping , unavailability of the required assay platform. 1 sample was received from Singapore, 0 from Egypt. No participant is analyzed, and no gene expression and CNV data is generated because the Affymetrix U133A GeneChip and SNPChip are unavailable. No participant will be analyzed, and no gene expression and CNV data will be generated in the future.
Arm/Group | Biology Samples-United States (US) | Biology Samples-Singapore | Biology Samples-Egypt
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Pattern and Frequency of XLP Gene Mutations Presenting With B-cell Lymphomas in the United States and Selected Geographic Regions
Description: Frequency of XLP mutation among boys will be calculated in each geographical region as well as in all regions pooled. The frequency is reported here as the number of boys with XLP gene mutations found in B-cell lymphomas boys.
Time Frame: 1 year after the participant enrollment
Population: We cannot obtain samples from other countries; thus cannot evaluate this objective, due to the PI leaving, difficulties caused by COVID-19, and, most importantly, changes in regulations on sending tumor material from institutions in other countries. We received 1 sample from Singapore and none from Egypt. For international sites, no clinical, laboratory or outcome features are available. Among US samples, 1 was tested XLP positive. No data was generated from the Singapore sample.
Measure: Count of Participants; unit: Participants
Groups:
- Biology Samples-United States (US): US Participants
- Biology Samples-Singapore: Singapore Participants
- Biology Samples-Egypt: Egypt Participants
Arm/Group | Biology Samples-United States (US) | Biology Samples-Singapore | Biology Samples-Egypt
Number analyzed (Participants) | 67 | 1 | 0
Participants | 1 | 0 | 0

5. Primary Outcome: Frequency of EBV Protein Expression (e.g., EBNA 3) in EBV-positive Lymphomas
Description: Frequency of EBV-positive BL will be calculated for each geographical region.
Time Frame: 1 year after the participant is enrolled
Population: We were unable to fully evaluate this measure due to PI leaving St. Jude, COVID-19 disruptions, and stricter regulations on sending tumor material from other countries. We received 5 participants at our institution and none showed EBV positivity. No sample was received from international sites. No EBV positivity test will be performed, and no further data will be generated in the future.
Measure: Count of Participants; unit: Participants
Arm/Group | Biology Samples-United States (US) | Biology Samples-Singapore | Biology Samples-Egypt
Number analyzed (Participants) | 5 | 0 | 0
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Overall Survival
Description: Overall survival (OS) will be estimated among eligible patients treated at SJCRH by the Kaplan-Meier estimator.
Time Frame: Up to 5 years after completion of therapy
Population: The study objective requires to obtain and analyze long-term outcome (OS and EFS) and toxicities in Groups A, B, C only. Patients in the "Biology Only" group only provide samples and are not treated on this protocol. Therefore EFS, OS and toxicities are only analysed and reported for Groups A, B and C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 86 | 22
percentage of participants | 100 [100 to 100] | 98.0 [86.4 to 99.7] | 94.7 [68.1 to 99.3]
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; Test type: Superiority; p = 0.5550, Log Rank

7. Other Pre Specified Outcome: Event-free Survival
Description: Event-free survival (EFS) will be estimated among eligible patients treated at SJCRH by the Kaplan-Meier estimator. The events will include: (1) death while in continuous CR, (2) relapse, (3) secondary malignancy, and (4) failure to achieve complete response (CR).
Time Frame: Up to 5 years after completion of therapy
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 86 | 22
percentage of participants | 100 [100 to 100] | 90.6 [82.0 to 95.2] | 81.8 [58.5 to 92.8]
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; Test type: Superiority; p = 0.3605, Log Rank

8. Other Pre Specified Outcome: Complete Response Rate
Description: Complete response rate will be estimated with exact 95% CI based on the binomial distribution, and it will be reported as the percentage of patients who reached complete remission among eligible patients treated at SJCRH
Time Frame: Up to 5 years after completion of therapy
Population: Only the 89 patients treated at St. Jude Children's Hospital are included in this analysis.The study objective requires to obtain and analyze long-term outcome (OS and EFS) and toxicities in Groups A, B, C only. Patients in the "Biology Only" group only provide samples and are not treated on this protocol. Therefore EFS, OS and toxicities are only analysed and reported for Groups A, B and C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 1 | 71 | 17
percentage of participants | 100 [2.5 to 100] | 90.14 [80.74 to 95.94] | 82.35 [56.57 to 96.20]
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C; Test type: Superiority; p = 0.6181, Chi-squared

ADVERSE EVENTS:
Time Frame: Acute adverse events were collected from each participant's on-study date through the end of therapy, through study completion, an average of 8 months. The timeframe for All-Cause Mortality is from start of therapy up to 5 years after completion of therapy.
Description: The "unknown risk patient" was consented and died prior to risk assignment or starting therapy. No additional adverse event data was captured.
  The "Biology Only" group only provide samples and were not treated on this protocol. No adverse event data was captured on these participants.
Arm/Group | Group A | Group B | Group C | Unknown Risk
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/86 | 1/22 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/86 | 0/22 | 0/0
Other Adverse Events (participants affected / at risk) | 3/5 | 77/86 | 21/22 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=5) | Group B (N=86) | Group C (N=22) | Unknown Risk (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 58 | 18 | NA
Mucositis oral (Gastrointestinal disorders) | 0 | 36 | 17 | NA
Enterocolitis infectious (Infections and infestations) | 0 | 13 | 8 | NA
Infections and infestations - Other, specify (Infections and infestations) | 0 | 9 | 6 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 8 | 5 | NA
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 8 | 5 | NA
Mucosal infection (Infections and infestations) | 0 | 7 | 7 | NA
Lung infection (Infections and infestations) | 0 | 7 | 4 | NA
Hypertension (Vascular disorders) | 0 | 7 | 3 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 5 | NA
Upper respiratory infection (Infections and infestations) | 0 | 6 | 3 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | NA
Thromboembolic event (Vascular disorders) | 0 | 6 | 0 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5 | 5 | NA
Colitis (Gastrointestinal disorders) | 0 | 5 | 5 | NA
Anemia (Blood and lymphatic system disorders) | 0 | 5 | 3 | NA
Fever (General disorders) | 0 | 5 | 3 | NA
Skin infection (Infections and infestations) | 0 | 5 | 3 | NA
Headache (Nervous system disorders) | 0 | 5 | 0 | NA
Sepsis (Infections and infestations) | 0 | 4 | 6 | NA
Hypotension (Vascular disorders) | 0 | 4 | 5 | NA
Alanine aminotransferase increased (Investigations) | 0 | 4 | 4 | NA
Neutrophil count decreased (Investigations) | 0 | 4 | 3 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | NA
Allergic reaction (Immune system disorders) | 0 | 4 | 3 | NA
Platelet count decreased (Investigations) | 0 | 4 | 2 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 2 | NA
Anal mucositis (Gastrointestinal disorders) | 0 | 4 | 0 | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 4 | NA
White blood cell decreased (Investigations) | 0 | 3 | 3 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | NA
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | NA
Oral pain (Gastrointestinal disorders) | 0 | 3 | 3 | NA
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 2 | NA
Lymphocyte count decreased (Investigations) | 0 | 2 | 4 | NA
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 4 | NA
Catheter related infection (Infections and infestations) | 0 | 2 | 2 | NA
Sinusitis (Infections and infestations) | 0 | 2 | 2 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | NA
Blood bilirubin increased (Investigations) | 0 | 1 | 3 | NA
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 2 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT01046825/Prot_SAP_000.pdf